CLINICAL TRIAL: NCT04745273
Title: The Effect of Ondansetron on the Efficacy of Tramadol
Brief Title: Interaction Between Tramadol and Ondansetron
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Sevgi Bilgen, Associate professor, Acibadem University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: SevgiB
Record Dates: First submitted 2021-01-31; First posted 2021-02-09 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cholecystectomy, Laparoscopic
Keywords: tramadol; ondansetron
MeSH Terms: interventions — Ondansetron

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ondansetron (Active Comparator): Participants will receive Kemoset 4 mg iv intraoperatively
  Interventions: Drug: Ondansetron 4 MG (Kemoset 4mg)
- Salin solution (Placebo Comparator): Participants will receive Salin solution 2ml (iv) intraoperatively
  Interventions: Other: Salin solution

INTERVENTIONS:
Drug: Ondansetron 4 MG (Kemoset 4mg) — Ondansetron 4mg (iv) will administer to participants
  Other Names: Kemoset
  Arms: Ondansetron
Other: Salin solution — Salin solution 2ml (iv) will administer to participants
  Arms: Salin solution

SUMMARY:
In the postoperative period; pain, nausea, and vomiting are undesirable side effects that reduce the patient's comfort and may lead to various complications. Ondansetron is frequently used as an antiemetic and tramadol hydrochloride is used for postoperative analgesia in laparoscopic cholecystectomy. However, some studies have reported that there is a drug interaction between these two drugs and they reduce each other's effects, thus requiring more analgesics in the postoperative period.

The aim of this study is; To evaluate whether ondansetron reduces the analgesic efficacy of tramadol hydrochloride in laparoscopic cholecystectomies.

DETAILED DESCRIPTION:
During the operation, 4 mg iv ondansetron (2mL) will be administered to the ondansetron group and 2mL iv 09% saline will be administered to the placebo group. The patients' heart rate, blood pressure, oxygen saturation, sedation score (with Ramsey Seading Score), amount of pain (with NRS), degree of nausea (with NRS), whether there is vomiting, whether analgesic or antiemetic treatment is required, and the amount of tramadol use will be recorded at 1, 2, 4, 8, 12 and 24 hours in the postoperative period.

ELIGIBILITY:
Inclusion Criteria:

60 patients over the age of 18, ASA I-II, undergoing laparoscopic cholecystectomy

Exclusion Criteria:

1. Patients under 18 years of age
2. Patients with known allergies to the drugs to be used
3. Pregnant and breastfeeding mothers
4. Patients who received antiemetic or cortisone within 24 hours before surgery
5. Patients with mental illness or epilepsy
6. Patients with alcohol or substance abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-09-02 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Interaction | 24 hours
  The hypothesis of this study is that if ondanstron is given together with tramadol peroperatively, tramadol consumption is increase postoperatively due to tramadol ondansetron interaction. The primary outcome measure is consumption of tramadol postoperatively for 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Bilgen, Assoc. Prof., Study Chair — Anethesiologist
Locations (1):
- Acibadem Kozyatagi Hastanesi, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Bilgen S, Erdogan Ari D, Ozveri E. The Effect of Ondansetron on the Analgesic Efficacy of Tramadol in Patients Undergoing Laparoscopic Cholecystectomy. Int J Clin Pract. 2022 Mar 8;2022:7387600. doi: 10.1155/2022/7387600. eCollection 2022. PMID 35685538